CLINICAL TRIAL: NCT05760443
Title: Mental Health Intervention Research in At-Risk Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4219
Record Dates: First submitted 2023-02-15; First posted 2023-03-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based intervention (Experimental): 6 week group mindfulness-based intervention
  Interventions: Behavioral: Learning to BREATHE

INTERVENTIONS:
Behavioral: Learning to BREATHE — Learning 2 BREATHE (L2B) is an empirically-supported, manualized mindfulness-based group program (Broderick, 2021). Participants attend 6 sessions of approximately 1.5 hours per session. "BREATHE" is an acronym: Body, Reflections, Emotions, Attention, Tenderness, Habits, Empowerment; each week's lesson is centered around one of the letters (week 1 encompasses both Body and the overall theme of the sessions, Empowerment). Sample activities of L2B include psycho-education on emotion and self-regulation, body scanning, sitting meditation, non-aerobic yoga, and walking meditation, designed to promote moment-to-moment awareness of mind-body experiences. In between sessions, participants are encouraged to practice brief mindfulness skills in their daily lives and to complete the "homework" assignments, such as an audio-guided body scan. Participants will have access to home-practice audio-recordings and will be queried about their completion of home-practice assignments.

SUMMARY:
The goal of the proposed research is to support adolescent health through providing inclusive evidence-based programming that is in line with community needs. Specifically, the investigators aim to: 1) investigate the effects of mindfulness-based intervention (MBI) on adolescent mental health, 2) identify underlying mechanisms (e.g., engagement, stress physiology, emotion regulation) of MBI for adolescent health and wellbeing 3) identify facilitators and barriers of engagement in MBI for community adolescents.

DETAILED DESCRIPTION:
Experiencing mental health problems during adolescence is associated with symptom worsening and recurrence later in life, as well as poorer physical health and increased risk for preventable chronic diseases. Mindfulness-based intervention (MBI) has been shown to support key skills and capacities that may protect against mental health challenges, including emotion regulation and stress physiology. Yet, MBI effects on health and wellbeing outcomes in adolescents are generally small and inconsistent across studies. This research will provide an opportunity for testing MBI in community adolescent samples, with a focus on clarifying underlying mechanisms and understanding subjective facilitators and barriers to engagement in MBI is critical.

In research with adolescents, L2B has been associated with improvements in emotion regulation and indicators of mental and physical wellbeing. In our previous work, the investigators delivered L2B as part of a broader healthy lifestyle program for families, and it was feasible and acceptable to adolescent participants. Delivering L2B is also consistent with the results of the 2020 Larimer County Needs Assessment, in which 48% of respondents indicated a need for more resources to support mental health and stress management for youth. Thus, given the solid evidence base for the benefits of L2B for adolescents, our experience delivering L2B to Northern Colorado teens in a previous phase of this community-engaged work, and the identified community need for inclusive, evidence-based mental health prevention programming for adolescents, the investigators will begin delivering L2B and evaluating the program's benefits on adolescent health and wellbeing.

The capacity of mindfulness, or present-centered, nonjudgmental attention, has also been associated with fewer mental health concerns in adolescents. However, meta-analyses and recent large-scale randomized controlled trials indicate that MBI does not always produce the desired outcomes in adolescents. This heterogeneity of findings indicates the need for mechanistic studies that closely examine the processes occurring during and between intervention sessions. This project both addresses an identified community need (inclusive mental health programming for adolescents) and will advance our understanding of the mechanisms that underlie MBI efficacy for supporting youth mental health in nonclinical samples.

This study will be a single-arm trial of an MBI utilizing a repeated measures assessment design. The single-arm nature keeps the project aligned with our goal of meeting community needs, and the multiple assessment timepoints (baseline, weekly across the 6-week intervention, follow-up) allows us to examine temporal ordering of changes in hypothesized mechanisms. With this project the investigators seek to elucidate the underlying mechanisms of mindfulness-based intervention effectiveness for adolescent health.

ELIGIBILITY:
Inclusion Criteria:

1) between the ages of 12-18 years old,

- 2) Reside in Larimer County or the surrounding area.

Exclusion Criteria:

* Adolescents will not take part in the program if they demonstrate active suicidal ideation and/or behavior.
* Adolescents will not take part in the program and/or research activities if they have a medical and/or psychological/behavioral condition that, in the opinion of the research team, could interfere with safety for themselves or others or interfere with the capability of the youth or other participants to potentially benefit from the program (e.g., severe emotional-behavioral disturbance, inability to follow facilitator directions) .

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation - Adolescent Report | 6 weeks
  Adolescent self-report on Difficulties in Emotion Regulation Scale - Short Form; The scale yields a sum score from 0-90 on 18 items. Higher scores indicate more difficulties in emotion regulation
Emotion Regulation - Parent Report | 6 weeks
  Parent self-report on Difficulties in Emotion Regulation Scale - Parent Version; The scale yields a sum score from 0-145 on 29 items. Higher scores indicate more difficulties in emotion regulation
Mindfulness - Attention | 6 weeks
  Adolescent self report on the Mindful Attention Awareness Scale; The scale yields a sum score from 0-75 on 15 items, and then an average will be taken. Higher scores reflect higher levels of dispositional mindfulness.
Mindfulness - Self Compassion | 6 weeks
  Adolescent self report on the Self Compassion Scale - Short Form; The scale yields a sum score from 0-60 on 12 items, and then an average will be taken. Higher scores reflect higher levels of self compassion.
Mindfulness - Behavioral Task | 6 weeks
  Adolescent will complete the Breath Counting Task, a 20-minute computer-administered objective measure of mindfulness. In the task, participants are required to count their breaths in cycles of nine, indicating each breath with a button press. Counting accuracy is calculated as 100% - (# of incorrect ongoing 9-counts + # of self-caught miscounts)/(# of ongoing 9-counts + # of self-caught miscounts).
Stress Reactivity - Respiratory Sinus Arrythmia | 6 weeks
  Respiratory changes will be measured measured by recording the rate and depth of the breathing cycle using a pneumograph transducer fastened around the center of the chest; this transducer measures changes in chest expansion and contraction. This data will be collected throughout a brief baseline period, a stressor task (the Trier Social Stress Task), and a recovery period.
Stress Reactivity - Skin Conductance | 6 weeks
  Skin conductance level will be measured by attaching two electrodes to the participant's fingertips (on the index and middle finger of the left hand). This data will be collected throughout a brief baseline period, a stressor task (the Trier Social Stress Task), and a recovery period.
Stress Reactivity - Heart Rate | 6 weeks
  Electrocardiogram (ECG) will be used to record the electrical signal of the heart using electrodes on both legs above the ankle both and above the right wrist. This will be collected throughout a brief baseline period, a stressor task (the Trier Social Stress Task), and a recovery period.
Stress Reactivity - Blood Pressure | 6 weeks
  A Dinamap Pro will be used to measure systolic and diastolic blood pressure. This will be collected throughout a brief baseline period, a stressor task (the Trier Social Stress Task), and a recovery period.
Mental health - Anxiety | 6 weeks
  Self report on Patient Reported Outcome Measurement Information System Emotional Distress Scale - Anxiety. The scale produces a sum score of 13 to 65 with higher scores indicating greater severity of anxiety.
Mental health - Depression | 6 weeks
  Self report on Patient Reported Outcome Measurement Information System Emotional Distress Scale - Depression. The scale produces a sum score of 14 to 70 with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Compassion for others | 6 weeks
  Self report on Compassion Scale. The scale yields a sum score from 5-80 with higher scores indicating more compassion for others
Stress appraisal | 6 weeks
  Self report on the Perceived Stress Scale. The scale yields sum scores on the PSS from 0 to 40 with higher scores indicating higher perceived stress.
Social Media Use | 6 weeks
  Self report on the Bergen Social Media Addiction Scale. The total score of Bergen Social Media Addiction Scale ranges from 6-30, with higher scores indicating more addictive tendencies in social media use.
Eating behavior | 6 weeks
  Self report on the Reward Based Eating Drive Scale. Items are summed for a total score between 5 and 45, with higher scores indicating more tendency toward reward-based eating.
Objectified Body Consciousness | 6 weeks
  Self report on the Body Surveillance and Body Shame subscales of the Objectified Body Consciousness Scale. Each scale contains 8 items. A sum score between 7 and 112 will be calculated, with higher scores indicating higher body consciousness.
Intervention liking and acceptability | 6 week follow up only
  Author-developed self report questions. Items will be on a scale of 1 to 5, with higher scores indicating greater liking of the program. Total possible scores will range from 5 to 25.
Engagement - Cognitive Behavioral | 6 weeks
  Adolescents will report on the 16-item Activity Engagement Scale. Sum scores are derived, with possible scores from 5 to 80, with higher scores indicating greater engagement.
Engagement - Value | 6 weeks
  Adolescents will complete the 7-item value subscale of the Intrinsic Motivation Inventory. Scores range from 7 to 49, with higher scores indicating more value motivation.
Engagement - Interest | 6 weeks
  Adolescents will complete the 7-item value subscale and the 7-item interest subscale of the Intrinsic Motivation Inventory. Scores range from 7 to 49, with higher scores indicating more interest motivation.
  the 8-item Teacher and Classmate Support Scale. They will also report on their home practice of mindfulness and complete the 15-item Applied Mindfulness Process Scale, which assesses the degree to which participants are applying mindfulness as discussed/trained in the intervention sessions. Observational assessments of engagement will be completed by outside raters.
Engagement - Teacher and Classmate Support | 6 weeks
  Adolescents will complete the 8-item Teacher and Classmate Support Scale. A sum score between 5 and 40 is derived, with higher scores indicative of more perceived support.
Engagement - Mindfulness | 6 weeks
  Adolescents will complete the 15-item Applied Mindfulness Process Scale, which assesses the degree to which participants are applying mindfulness as discussed/trained in the program. A sum all 15 items yields score ranging from 0-60, with higher scores indicating more application of mindfulness
Engagement - Observational | 6 weeks
  Independent observers will code videotaped sessions of mindfulness training using the Engagement Observation Protocol. Scores range from 3 to 15, with higher scores indicating more engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Shomaker, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No